CLINICAL TRIAL: NCT01004276
Title: A Cluster Randomized Controlled Pilot Trial of the Effect of a New, Improved Smoking Cessation Management Module, Compared With Use of the Standard Version of Such a Management Module, on Smoking Counselling Initiation and Continuation Rates in Primary Care Practices Currently Using P-PROMPT Chronic Disease Management System in Ontario
Brief Title: Increasing Smoking Cessation Counselling in Primary Care Using a Chronic Disease Management System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: McMaster University (Other)
Collaborators: Centre for Addiction and Mental Health (Other)
Responsible Party: Natalie T. MacLeod, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 09-341
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Last update posted 2009-10-29 (Estimated); Status verified 2009-10

CONDITIONS: Delivery of Health Care; Smoking Cessation
Keywords: primary health care; delivery of health care; smoking cessation; chronic disease; disease management; pilot projects
MeSH Terms: conditions — Smoking Cessation; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Improved module (Experimental)
  Interventions: Other: New, improved smoking cessation management module
- Standard module (No Intervention)

INTERVENTIONS:
Other: New, improved smoking cessation management module — The intervention that will be tested is an improved smoking cessation management module in an existing chronic disease management system, P-PROMPT CDMS. This module includes the following components: a) the Patient Care Status and Update Form, b) the smoking registry and c) patient prompts.
  Arms: Improved module

SUMMARY:
This pilot study will determine the feasibility of studying a new smoking cessation management module in an existing chronic disease management system. The new module is intended to help healthcare providers deliver more smoking cessation counselling to their patients.

ELIGIBILITY:
Inclusion Criteria:

* Physician subscribers to P-PROMPT CDMS

Exclusion Criteria:

* Paper users
* Physicians expected to retire during the course of the study
* Physicians whose billing files are not set-up with DataSynch

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Smoker Identifying Cards | 3 months post-intervention
Chronic disease management system's activity log | monthly post-intervention

SECONDARY OUTCOMES:
Smoking cessation counselling billing codes from physician's remittance advice files | monthly post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Natalie T. MacLeod, M.Sc. Candidate, Principal Investigator — McMaster University; Rolf J. Sebaldt, MD, Principal Investigator — McMaster University; Peter Selby, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (2):
- Canada (2):
  - McMaster University, Hamilton, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario